CLINICAL TRIAL: NCT02445859
Title: Colo-Pro Pilot: A Pilot Study to Compare Standard Single Dose Antibiotic Prophylaxis to Bolus-continuous Infusion Dosed Antibiotic Prophylaxis for the Prevention of Infections After Colorectal Surgery
Brief Title: Continuous Antibiotic Prophylaxis in Colorectal Surgery
Acronym: Colo-Pro
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Andrew Kirby, Associate clinical professor, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MB15/130
Record Dates: First submitted 2015-05-13; First posted 2015-05-15 (Estimated); Results first posted 2019-09-12 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Surgical Site Infection
Keywords: Antibiotic; prophylaxis; surgical site infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard regimen (Active Comparator): Cefuroxime 1.5grams pre-operatively Repeated every 4 hours
  Interventions: Drug: Cefuroxime 4 hourly bolus
- Interventional regimen (Experimental): Cefuroxime continuous infusion targeting 64mg/l serum concentrations.
  Interventions: Drug: Cefuroxime 4 hourly bolus

INTERVENTIONS:
Drug: Cefuroxime 4 hourly bolus — Cefuroxime loading dose followed by a continuous infusion dosed according to renal function. Dosed to target a serum concentration of 64mg/L.

SUMMARY:
We propose to randomise patients due to undergo colorectal surgery to standard antibiotic prophylaxis or an interventional antibiotic prophylaxis regimen and assess surgical wound infection rates. Standard antibiotic prophylaxis is a pre-operative injection of cefuroxime, repeated every 4 hours. The intervention regimen is a loading dose of cefuroxime followed by a continuous infusion of cefuroxime until the end of surgery. The intervention regimen dosing will be calculated using a patient's renal function and body weight. The intervention regimen will target a free serum drug concentration of 64mg/L. This serum level is 4x the MIC90 for colonising Enterobacteriaceae. The rational for this dosing regimen is summarised below. The primary objective of the study is to reduce by 50% the rate of surgical wound infections after colorectal surgery.

DETAILED DESCRIPTION:
An expert assessment is that fT>MIC is the measure most likely to be applicable to prophylaxis. But this measure is not achieved by standard prophylaxis regimens. Neither do clinical data suggest this target achieves optimal prophylaxis. Therefore there is an opportunity to optimise antibiotic prophylaxis dosing. As the exposure response-relationship (pharmacodynamic target) is unknown we could either complete a number of studies exploring different relationships, or compare standard treatment to a single regimen which included a number of exposure-response relationships. The two most common exposure-response relationships are the CMAX/MIC ratio and the fT>MIC. And it has been reported that killing, as opposed to inhibition used in MIC values, is optimised by achieving 4 times an MIC value. An antibiotic prophylaxis regimen which achieved drug concentrations of 4xMIC for the duration of surgery would therefore achieves a high CMAX/MIC ratio, high T>MIC, and optimise bacterial killing. Therefore, standard dose antibiotic prophylaxis will be compared against a PD target dosed antibiotic prophylaxis regimen. The PD target will be a free serum antibiotic concentration of 4xMIC90 for Enterobacteriaceae against cefuroxime. Continuous infusion of antibiotic prophylaxis will ensure there is continuous targeting of this drug level throughout the operation.

ELIGIBILITY:
Inclusion criteria

* Undergoing colorectal surgery (incision, excision or anastomosis of the large bowel, including anastomosis of small to large bowel)
* Age >18.
* Expected duration of surgery > 2hours
* Creatinine clearance > 40 ml/min
* Cefuroxime/metronidazole are appropriate antibiotic prophylaxis regimens.
* Patient capable of giving informed consent
* Patients undergoing colorectal surgery plus additional surgery e.g. plastic surgery, urological surgery, gynaecological surgery.
* If it is not possible to obtain intra-operative blood samples e.g. difficult vascular access, or pre-operative swabs e.g. anatomy makes it difficult to obtain, patients will be included and this information treated as missing data. Patients on antibiotic treatment for an existing infection (except SSIs) can be included in the study

Exclusion Criteria:

* Unable to consent
* Pregnancy
* Expected duration of surgery <2hours
* Creatinine clearance <40ml/min
* Individual level microbiological advice for non cefuroxime based prophylaxis
* Cephalosporin allergy
* Penicillin allergy (hypersensitivity reaction only)
* Coumarin (warfarin and acenocoumarol) treatment
* Active blood borne virus infection e.g. HIV, hepatitis.
* Seizure history
* Concurrent use of probenecid
* Current participation in a research project aimed at reducing SSIs
* Antibiotics for treatment of a systemic Gram negative infection within 2 hours of initiation of surgery (Vancomycin, Teicoplanin, Daptomycin, Linezolid, Flucloxacillin. Nitrofurantoin and Clarithromycin would be permissible antibiotics without systemic Gram negative antibiotics).
* A current diagnosis of a SSI at the time of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Kirby, Principal Investigator — The University of Leeds
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kirby A, Asin-Prieto E, Burns FA, Ewin D, Fatania K, Kailavasan M, Nisar S, Pericleous A, Troconiz IF, Burke D. Colo-Pro: a pilot randomised controlled trial to compare standard bolus-dosed cefuroxime prophylaxis to bolus-continuous infusion-dosed cefuroxime prophylaxis for the prevention of infections after colorectal surgery. Eur J Clin Microbiol Infect Dis. 2019 Feb;38(2):357-363. doi: 10.1007/s10096-018-3435-z. Epub 2018 Dec 5. PMID 30519893

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Regimen: Cefuroxime 1.5grams pre-operatively Repeated every 4 hours
  Cefuroxime bolus-continuous infusion: Cefuroxime 1.5 grams pre-operatively, repeated 4 hourly during surgery.
Period: Overall Study
Arm/Group | Standard Regimen | Interventional Regimen
Started | 45 | 45
Completed | 43 | 42
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Population: The analysis population was on an intention to treat basis
Groups:
- Standard Dosing: Intravenous (IV) cefuroxime 1.5g bolus administered four-hourly throughout surgery
- Intervention Dosing: Cefuroxime bolus-continuous dosing was based on targeting non-protein bound (free) serum concentrations of antibiotic at 64mg/L throughout surgery
- Total: Total of all reporting groups
Arm/Group | Standard Dosing | Intervention Dosing | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] — Collection by review of medical records
  years | 58 (17) | 61 (17) | 60 (17)
Sex: Female, Male [Count of Participants; unit: Participants] — Collection by review of medical records
  Participants
    Female | 24 | 27 | 51
    Male | 21 | 18 | 39
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With a Surgical Site Infection
Description: Superficial and deep surgical site infections as defined by the CDC (Centre's for Disease Control) definitions of surgical site infections.
Time Frame: Number of patients with a surgical site infection within 30 days of a colorectal surgical procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Regimen | Interventional Regimen
Number analyzed (Participants) | 43 | 42
Participants | 10 | 13

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Standard Regimen | Interventional Regimen
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/42
Serious Adverse Events (participants affected / at risk) | 3/43 | 5/42
Other Adverse Events (participants affected / at risk) | 0/43 | 0/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Regimen (N=43) | Interventional Regimen (N=42)
Anastomotic leak (Gastrointestinal disorders) | 0 (0) | 3 (3)
Unplanned surgical procedure (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastrointestinal bleed (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pleural effusion with pleural drain insertion (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Regimen (N=43) | Interventional Regimen (N=42)
Clostridium difficile infection (Gastrointestinal disorders) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
These patients are expected to have multiple adverse events. We only formally collected all serious adverse events, plus specific events e.g. C.difficile. As a pilot trial we have learned about the collection of adverse events in this patient group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-10-10): https://cdn.clinicaltrials.gov/large-docs/59/NCT02445859/Prot_SAP_000.pdf
  • Informed Consent Form (2015-11-24): https://cdn.clinicaltrials.gov/large-docs/59/NCT02445859/ICF_001.pdf